CLINICAL TRIAL: NCT06336798
Title: Effect of Pioglitazone on Mitochondrial Metabolism in Pulmonary Hypertension Due to Chronic Lung Disease
Brief Title: Bioenergetic Effect of Pioglitazone in CLD-PH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Aaron W Trammell, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005871; K23HL166775 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension; Pulmonary Hypertension Due to Lung Diseases
Keywords: Pulmonary Hypertension; Chronic Lung Disease; Pioglitazone
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pioglitazone, Then Placebo (Experimental): Participants will first receive a 30 mg tablet of Pioglitazone once daily for 28 days. After a washout period of 14 days, they will then receive a Placebo tablet (matching Pioglitazone 30 mg tablet) once daily for 28 days.
  Interventions: Drug: Pioglitazone 30mg; Drug: Placebo; Diagnostic Test: Labs
- Placebo, Then Pioglitazone (Experimental): Participants will first receive a Placebo for 28 days. After a washout period of 14 days, they will then receive a 30 mg Pioglitazone tablet once daily for 28 days.
  Interventions: Drug: Pioglitazone 30mg; Drug: Placebo; Diagnostic Test: Labs

INTERVENTIONS:
Drug: Pioglitazone 30mg — Study participants will take Pioglitazone 30 mg PO daily
  Other Names: Actos
Drug: Placebo — Study participants will take a placebo PO daily
Diagnostic Test: Labs — Labs will be performed for Urine HCG, Complete Blood count (CBC), Chemistry Panel, Fasting lipids, insulin, glucose, and Bioenergetic analysis (platelets).
  Other Names: Diagnostic labs

SUMMARY:
The goal of this clinical trial is to learn about the safety and efficacy of Pioglitazone in people with Pulmonary Hypertension (PH) due to Chronic Lung Disease (CLD). The main question it aims to answer is:

• Whether pioglitazone affects mitochondrial oxygen utilization in patients with PH due to CLD.

Participants will be asked to take pioglitazone or placebo once daily for 28 days followed by a washout period of 2 weeks followed by 28 days of the other study drug (participants randomized to placebo followed by pioglitazone or pioglitazone followed by placebo).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a state of chronic elevated pressure in the pulmonary circulation. PH has multiple possible causes, clinically classified into 5 separate groups according to the World Symposium on PH classification scheme. PH is common in adults, with increasing prevalence with age, and is associated with significant symptom burden and mortality. In the U.S., approximately 1.5 million U.S. adults have PH, including 5-10% of people >65.

Metabolic abnormalities have been highlighted recently as contributing to PH pathogenesis, disease severity, and outcome. In pre-clinical studies, reduced mitochondrial metabolism (oxidative phosphorylation) and reliance on alternative metabolic pathways (glycolysis) have been shown to promote pulmonary vascular remodeling and PH. Mechanistic investigation has shown that reduced PPARγ activity in lung vascular cells is necessary and sufficient to cause cellular proliferation and dysfunction followed by PH, all of which can be reversed by available pharmacotherapies designed to activate PPARγ.

Metabolic changes have been demonstrated in 1) lung vessels from multiple PH animal models and 2) humans with PAH 3) right ventricle from humans with PAH, 4) skeletal muscle from humans with PAH, 5) circulating platelets from humans with PAH and PH due to left heart disease. Clinical trials of therapies that activate PPARγ have not been previously conducted in patients with PH but are believed by experts in the field to be a highly promising therapeutic approach.

In this trial, the investigators will study the mitochondrial metabolic effects ("bioenergetics") of pioglitazone, an available medication from the class of thiazolidinedione (TZD) drugs that activate PPARγ. This medication is FDA-approved for the treatment of Type II diabetes mellitus (DM). Pioglitazone has been studied in non-diabetics with diverse other conditions demonstrating safety.

The study team will assess cellular energy metabolism through a sophisticated assay of bioenergetics. The investigators and others have shown that bioenergetics can be measured in isolated platelets obtained from a peripheral blood draw in patients with PH and other diseases. Furthermore, others have shown that in PAH, platelet bioenergetics correlate with known disease-relevant metabolic changes in lung blood vessels. In this study, the team will assess the effect of pioglitazone on bioenergetic parameters in platelets isolated from whole blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent form
* Stated willingness to comply with all study procedures for the duration of the study
* Confirmed to have pulmonary hypertension (PH) due to chronic lung disease at screening

  * Pulmonary hypertension is defined based on meeting all three of the following measured at rest during the RHC:

    * Mean pulmonary artery pressure >20 mmHg
    * Pulmonary artery wedge pressure ≤15 mmHg
    * Pulmonary vascular resistance > 2 Wood units
  * Pulmonary hypertension is classified in Group 3: PH associated with lung diseases and/or hypoxia
* Medications approved for the treatment of pulmonary hypertension must be at a stable dose for at least 30 days
* Ability to take oral medication and be willing to adhere to the study intervention regimen
* For females of reproductive potential: agreement to use highly effective contraception during study participation and for an additional 4 weeks after the end of study participation.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with a partner
* Agreement to adhere to Lifestyle Considerations (below) throughout the study duration o During this study, participants are asked to arrive in the clinic for study visits in the fasting state. Specifically, participants should abstain from any caloric intake for 6 hours before arrival for the study visit.

Exclusion Criteria:

* Diabetes mellitus (type 1 or type 2), present within the preceding 1 year
* Personal history of symptomatic hypoglycemia within 90 days preceding enrollment
* Personal outpatient use of pioglitazone, rosiglitazone, metformin, insulin, or other medications for the indication of diabetes within 90 days preceding enrollment
* History of left ventricular failure (systolic or diastolic)
* Pulmonary hypertension due to Group 2 PH (PH due to left heart disease)
* History of prior or active bladder cancer
* Thrombocytopenia (diagnosis or known platelet count ≤120) within 90 days preceding enrollment
* Platelet count ≤120 during screening or on the day of enrollment hypertension due to chronic lung disease
* Cystic fibrosis
* Pregnancy or lactation
* Current tobacco use
* Known allergic reaction to components of the study medication (pioglitazone)
* Treatment with another investigational drug within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in Mitochondrial metabolism parameters: Spare respiratory capacity | Day 1, Day 28, Day 70
  Mitochondrial metabolism is measured using a research protocol employing the Agilent Seahorse extracellular flux bioanalyzer. Standard Seahorse assay protocols have been adapted for use with human platelets .
  Spare respiratory capacity (SRC) is calculated by (maximal respiration) - (basal respiration) during the mitochondrial stress test. The value is reported in pmol/min.
Change in Mitochondrial metabolism parameters: Maximal respiration | Day 1, Day 28, Day 70
  Maximal Respiration is calculated by: (post-carbonyl cyanide 4-(trifluoromethoxy) phenylhydrazone(FCCP) - (nonmitochondrial respiration) during the mitochondrial stress test. The value is reported in pmol/min.
Change in Mitochondrial metabolism parameters: Basal respiration | Day 1, Day 28, Day 70
  Basal respiration is calculated by (Baseline) - (nonmitochondrial respiration) ) during the mitochondrial stress test. The value is reported in pmol/min.

SECONDARY OUTCOMES:
Number of hypoglycemia incidences | Day 1, Day 28, Day 70
  Participants experiencing symptoms of hypoglycemia will be identified and reported.
Number of participants with leg edema | Day 1, Day 28, Day 70
  Participants reporting edema (>2) will be captured.
Change in BNP levels | Day 1, Day 28, Day 70
  Change in Brain Natriuretic Peptide from the baseline will be calculated. Unit is pg/ml
Change in Six minute walk distance (6MWT) | Day 1, Day 28, Day 70
  The six-minute walk test (6MWT) is a standardized test of exercise capacity commonly used in patients with heart failure, lung disease, PH, and in pre-lung transplant evaluation. Results will be recorded as the distance walked in meters.
Change in Borg dyspnea score | Day 1, Day 28, Day 70
  Borg dyspnea score assessed before and after 6MWT. The Borg dyspnea score is a rating of dyspnea that is scored between 0 and 10. Higher scores indicate worse dyspnea.
Change in NYHA/WHO Functional Classification | Day 1, Day 28, Day 70
  The New York Heart Association / World Health Organization Functional Classification (NYHA/WHO FC) is a symptom-based score graded on a scale from I-IV. It is used to objectively assess severity of symptoms for patients with heart failure, PH, and other cardiopulmonary conditions. In this study, NYHA/WHO FC will be recorded at each study visit. Higher scores indicate a higher degree of functional limitation.
Change in University of California San Diego Shortness of Breath Questionnaire score | Day 1, Day 28, Day 70
  The University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) is a 24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living. It is self-completed by participants and is validated in multiple languages (including US English) and in diseases including COPD, ILD, and general states of dyspnea. Each of the 24 items is scored on a six-point scale (0-5). Total scores range from 0 to 120 with higher scores indicating worse dyspnea.
Change in emPHasis-10 Questionnaire score | Day 1, Day 28, Day 70
  The emPHasis-10 questionnaire consists of 10 items that address breathlessness, fatigue, control, and confidence and is designed to assess the impacts that PH has on a person's quality of life. Each of the items is scored on a six-point scale (0-5). emPHasis-10 scores range from 0 to 50 with higher scores indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Trammell, Principal Investigator — Emory University
Locations (1):
- Emory Healthcare System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No